CLINICAL TRIAL: NCT06018688
Title: A Phase II Study Evaluating Osimertinib Combined With Aspirin Neoadjuvant Therapy for Resectable EGFR Mutated Non-small Cell Lung Cancer (NSCLC)
Brief Title: Osimertinib Combined With Aspirin Neoadjuvant Therapy for Resectable EGFR Mutated NSCLC Patients.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Yong He, Professor, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEWCOAST
Record Dates: First submitted 2023-08-04; First posted 2023-08-31 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Non Small Cell Lung Cancer; EGFR Gene Mutation
Keywords: Non-Small Cell Lung Cancer; Aspirin; Osimertinib; EGFR-TKI; neoadjuvant therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib; Aspirin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- osimertinib and aspirin (Experimental): Osimertinib and Aspirin starting at a dose of 80 mg and 100mg once a day, orally with meals.The participants will undergo a two-month combination therapy, unless there is tumor progression (worsening) or intolerable toxic reactions that necessitate early termination of the drug treatment. Aspirin will be discontinued one week prior to the surgery.
  Interventions: Drug: Osimertinib; Drug: Aspirin

INTERVENTIONS:
Drug: Osimertinib — Osimertinib is a 3rd-generation EGFR-TKI used to treat NSCLC patients with resistance to 1st generation EGFR-TKI due to T790M mutation. It has been approved in clinical applications by the FDA in 2015.
  Other Names: OSI
Drug: Aspirin — Aspirin, also known as acetylsalicylic acid (ASA), is a verysafe medication used to treat pain,fever, or inflammation.
  Other Names: ASP

SUMMARY:
This is a single-center, prospective, single-arm, phase II study of Osimertinib combined with Aspirin neoadjuvant therapy for resectable, EGFR mutated non-small cell lung cancer (NSCLC). It is mainly aimed at the population of patients with primary IIA- IIIA EGFR sensitive mutations that are intended to be treated with Osimertinib neoadjuvant therapy.

DETAILED DESCRIPTION:
Lung cancer is currently the leading cause of cancer-related deaths in humans, with its incidence and mortality rates continuously rising. Among them, non-small cell lung cancer (NSCLC) accounts for the vast majority of lung cancer cases (approximately 80%). About one-third of NSCLC cases are early-stage and potentially resectable. Curative surgical resection is the primary treatment approach for these patients. However, even with curative surgery, the 5-year survival rate of patients still needs improvement. It has been reported that approximately 30-55% of early-stage NSCLC patients experience recurrence within 5 years after surgery, indicating the presence of occult micro-metastases in early NSCLC. Neoadjuvant therapy before surgery can eliminate micro-metastases, downsize tumors, and reduce the risk of recurrence, thereby improving patient prognosis and extending survival. Previous studies have shown that neoadjuvant chemotherapy only achieves a 5% improvement in overall survival (OS) for patients, and the toxic side effects of chemotherapy limit its broad clinical application. Therefore, there is an urgent need for better neoadjuvant treatment strategies to enhance patient survival.

Research has shown that the epidermal growth factor receptor (EGFR) plays a significant role in the occurrence and progression of non-small cell lung cancer (NSCLC). For resectable stage IIA to IIIB NSCLC patients without EGFR mutations, the emergence of neoadjuvant immunotherapy combined with chemotherapy has been found to significantly prolong the patient's progression-free survival, improve the pathological complete response rate (pCR), and not increase the incidence of adverse events, thus providing survival benefits to patients. In the case of resectable stage IIA to IIIB NSCLC patients with EGFR mutations, several targeted neoadjuvant treatment attempts using third-generation EGFR-TKIs like osimertinib have been made, with promising data demonstrating favorable outcomes.

The 2019 World Conference on Lung Cancer (WCLC) reported a phase II clinical study using osimertinib as neoadjuvant therapy for patients with EGFR mutant NSCLC. Twenty-seven patients with stage I-IIIA EGFR mutant NSCLC received 1-2 months of osimertinib as neoadjuvant treatment prior to surgery. The major pathological response rate (MPR) for 6 assessable patients was 16%, and the objective response rate (ORR) was 66%. Thirty-three percent of patients achieved pathological downstaging. In an updated efficacy evaluation of 27 patients presented at the 2023 American Society of Clinical Oncology (ASCO) meeting, the MPR was 15%, ORR was 48%, R0 resection rate was 89%, median disease-free survival (mDFS) was 32.4 months, and median overall survival (mOS) was not reached. Another real-world retrospective study presented at the 2021 WCLC also explored the efficacy and safety of osimertinib in neoadjuvant therapy for stage I-IIIB patients. Seventeen patients who received osimertinib as neoadjuvant treatment had an MPR of 23.5%, pathological complete response (pCR) rate of 5.9%, and ORR of 88.2%. Overall, the treatment was well-tolerated. The mid-term results of the NEOS study presented at the 2021 ASCO Annual Meeting further confirmed the benefits of osimertinib as neoadjuvant therapy, although the data is still immature. From October 17, 2018, to June 8, 2021, a total of 88 patients were screened, and 40 patients were ultimately enrolled. Among the 38 patients who completed 6 weeks of osimertinib neoadjuvant therapy, the ORR was 71.1% , and the disease control rate reached 100%. This indicates that no disease progression occurred during the neoadjuvant treatment, and 71.1% of patients had significant tumor shrinkage, creating an opportunity to reduce the extent of surgical resection, decrease the difficulty of surgery, and improve surgical outcomes. However, among the 28 patients with assessable pathology, only 11% achieved MPR, and only 1 patient (4%) achieved pCR. It is well known that pathological response rates are closely related to postoperative recurrence and survival time. It would be clinically significant to further enhance the pathological response rate of osimertinib neoadjuvant patients through combination therapy strategies, which could reduce postoperative recurrence rates and improve overall survival.

Aspirin, a classic drug known for its antiplatelet effects, exhibits safety, affordability, and easy accessibility. Its potential role in cancer treatment has been widely explored. Recent studies have demonstrated the following:1. Women who take aspirin at least three times a week have a 16% reduced risk of developing breast cancer.2. Aspirin enhances the efficacy of the anti-tumor drug sorafenib in mouse models of lung cancer and melanoma with RAS gene mutations.3. By binding to the key amino acid Glu225, aspirin inhibits enzymatic activity of acetylheparinase, thereby suppressing tumor angiogenesis and metastasis.4. Aspirin boosts the effectiveness of T-cell therapy and enhances the body's immune response against cancer.5. Aspirin has received FDA approval for its preventive use in colorectal cancer.Numerous clinical and basic trials have validated the role of aspirin in cancer prevention and treatment. Moreover, our earlier research indicated that aspirin improves the immunosuppressive microenvironment associated with osimertinib, activates cytotoxic T-cell function, and enhances the killing ability of T cells against tumor cells, ultimately promoting tumor cell apoptosis. Lung cancer patients inherently experience a hypercoagulable state and are prone to critical cardiovascular events. Regular low-dose aspirin usage reduces the incidence of coronary events in lung cancer patients. Therefore, if further evidence confirms aspirin's ability to overcome osimertinib resistance beyond its antiplatelet effects, combining osimertinib with aspirin in neoadjuvant therapy for NSCLC patients could potentially enhance pathological response, reduce postoperative recurrence, and further improve the overall prognosis of patients eligible for surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with resectable stage IIA-IIIA lung adenocarcinoma.
2. Patients with EGFR sensitizing mutations (Ex19del or L858R).
3. Intended neoadjuvant therapy with osimertinib, with an anticipated survival expectancy of more than 3 months.
4. ECOG PS 0/1.
5. Primary lesion diameter of at least 1 cm.
6. Patients who have previously taken or are currently taking aspirin therapy are allowed.

Exclusion Criteria:

1. Currently receiving other anticoagulant therapy.
2. Previously treated with systemic therapy for NSCLC.
3. Other positive driver mutations, including ALK, ROS1, MET14 exon skipping, BRAF, RET, etc.
4. Contraindications to the use of osimertinib and aspirin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response | Within 1 month after surgery
  MPR refers to the percentage of residual viable tumor cells within the tumor bed after neoadjuvant treatment, with a threshold of ≤10%, regardless of the presence of residual viable tumor cells in the lymph nodes.

SECONDARY OUTCOMES:
Disease Free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months.
  DFS was defined as the time from complete surgical resection to recurrence or death due to any reason.
Objective Response Rate | 1 week before surgery
  Objective response rate (ORR) refers to the proportion of patients in a clinical trial or treatment setting whose tumor size reduces or disappears (partial or complete response) in response to the therapy being administered.
Disease Control Rate | 1 week before surgery
  Disease control rate (DCR) describes the percentage of patients with advanced cancer whose therapeutic intervention has led to a complete response, partial response, or stable disease.
Pathologic complete response | Within 1 month after surgery
  PCR refers to the absence of residual viable tumor cells in the tumor bed and lymph nodes after neoadjuvant therapy.

IPD SHARING:
Plan to Share IPD: Undecided